CLINICAL TRIAL: NCT07023016
Title: Comparative Assessment of Efficacy & Safety of Sacubitril/Valsartan Versus Ramipril in Patients With Renal Dysfunction Hospitalized With Acute Decompensated Heart Failure - CAESAR (a Randomized Controlled Trial)
Brief Title: Comparative Assessment of Efficacy & Safety of Sacubitril/Valsartan Versus Ramipril in Patients With Renal Dysfunction Hospitalized With Acute Decompensated Heart Failure
Acronym: CAESAR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Heart Institute, Egypt (Other Government)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Younis, Cardiology Researcher, National Heart Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD-464-2023
Record Dates: First submitted 2025-06-08; First posted 2025-06-15 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Acute Decompensated Heart Failure (ADHF); Chronic Kidney Disease (CKD)
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — sacubitril and valsartan sodium hydrate drug combination; Ramipril; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sacubitril / Valsartan (Experimental)
  Interventions: Drug: Sacubitril / Valsartan
- Ramipril (Active Comparator)
  Interventions: Drug: Ramipril (ACE-inhibitor)

INTERVENTIONS:
Drug: Sacubitril / Valsartan — Patients will receive sacubitril/valsartan at an initial dose of 24/26 mg Bid.
  Arms: Sacubitril / Valsartan
Drug: Ramipril (ACE-inhibitor) — Patients will receive ramipril at an initial dose of 2.5 mg Bid.
  Arms: Ramipril

SUMMARY:
Sacubitril/valsartan is an established medication for heart failure. However, data still lags in its use in heart failure patients with chronic kidney disease. Sacubitril/valsartan is manufacturer-labeled for use in patients with eGFR < 30 ml/min/1.73 m2 at an initial dose of 24/26mg twice daily. However, to the best of our knowledge, the concept of sacubitril/valsartan or ACEi in patients with chronic kidney disease & presenting with decompensated heart failure has not yet been explored fully.

ELIGIBILITY:
Inclusion Criteria: All the following should be met:

* Acute decompensated heart failure (ADHF)
* Left ventricular ejection fraction (LVEF) below 40%
* Renal dysfunction; defined as eGFR of 30mL/min/1.73m2 to less than 60mL/min/1.73m2 in relation to the level of urinary albumin/creatinine ratio (uACR) based on the 2024 Kidney Disease: Improving Global Outcomes (KDIGO) clinical practice guidelines for the evaluation and management of CKD.
* A minimum blood pressure (BP) ≥ 105/60 mmHg.
* Independent of any inotropic or vasopressor support in the previous 24 hours before inclusion and randomization.
* No more than 72 hours had passed since admission to the heart failure unit.
* Patients should have had a New York Heart Association (NYHA) functional class II-IV, in addition to symptoms of volume overload at the time of presentation to the emergency room.

Exclusion Criteria:

* Patients who were on sacubitril/valsartan or ACEI/ angiotensin receptor blocker (ARB) prior to inclusion.
* Patients with AKI on presentation OR in the last 3 months OR had ≥ 2 hospital admissions in the last 12 months for AKI.
* History of known or suspected hypersensitivity, contraindications, or intolerance to any of the study drugs including ACEI, ARB or sacubitril (neprilysin inhibitor).
* Requirement for double treatment with both ACEI and ARB.
* Serum potassium (K+) level ≥ 5.0 mmol/L at randomization.
* A recent major adverse cardiovascular/cerebrovascular event within 1 month (acute coronary syndrome, stroke, transient ischemic attack, etc.).
* Patients with hemodynamically significant primary valvular lesion.
* Known hepatic impairment with a model for end-stage liver disease (MELD) score >10. 23
* History of malignancy of any organ system within the past year with a life expectancy < 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Difference in mean eGFR (mL/min/1.73m2) between both groups at 12 weeks post-randomization. | 12 weeks

SECONDARY OUTCOMES:
Number of patients in each group who develop worsening renal function throughout the study period. | 12 weeks
  Defined as a 50% increase in the serum creatinine level (mg/dL) from baseline and/or a drop in eGFR by more than 25 ml/min/1.73m2.
Number of events in each group for hyperkalemia throughout the study period. | 12 weeks
  Defined as a rise in serum potassium level to ≥ 5.5 mEq/L .
Number of events in each group for symptomatic hypotension throughout the study period. | 12 weeks
  Defined as the subjective sense of dizziness or lightheadedness, blurred, or fading of vision, fainting, fatigue, difficulty concentrating and/or nausea in the presence of a BP of 90/60mmHg or lower.
Number of events in each group for angioedema throughout the study period. | 12 weeks
  Defined as a swelling (edema) of the dermis, subcutaneous tissue, mucosa, and submucosal tissues.
Difference between uACR levels (gm/mg) in each group at 12 weeks post-randomization. | 12 weeks
Difference between NT-proBNP levels (pg/mL) in each group at 12 weeks post-randomization | 12 weeks
Difference between LVEF (%) of each group at 12 weeks post-randomization | 12 weeks

OTHER OUTCOMES:
HF rehospitalization: this will include the total number of patients in each group who will require hospital re-admission for ADHF. | 12 weeks
All-cause mortality: this will include the total number of deaths in each group regardless of the underlying cause. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hesham Salah Eldin Taha, MD, Study Director — Cairo University; Omar Younis, Msc, Principal Investigator — National Heart Institiute, Cairo - Egypt
Locations (2):
- Egypt (2):
  - Cairo University Hospitals, Cairo
  - National Heart Institute, Cairo

IPD SHARING:
Plan to Share IPD: No